CLINICAL TRIAL: NCT07020715
Title: An Autologous and Antigen-specific Cell-based Therapy of Vitamin D3-treated and Myelin-derived Peptide Loaded Tolerogenic Dendritic Cells in Subjects With Progressive Forms of Multiple Sclerosis: a Phase IIa, Open-label, Self-controlled, Multi-center Clinical Trial
Brief Title: A Phase IIa Study of Vitamin D3 Tolerogenic Dendritic Cells (tolDC) for Multiple Sclerosis
Acronym: MS-tolDC_2a
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Fundació Institut Germans Trias i Pujol (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCRG22-002 / FWO-TBM T002523N; T002523N (Other Grant/Funding Number: FWO); 2025-522040-40-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-10

CONDITIONS: Multiple Sclerosis
Keywords: Tolerogenic dendritic cells; tolDC; Phase IIa; Multiple Sclerosis; MS; Patient Safety; Efficacy
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Participants will receive six administrations of the tolDC vaccine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intradermal Arm: tolerogenic dendritic cells (tolDC) (Experimental): Each vaccine (15x10E6cells in 500 µL solution with 5% human albumin supplemented with 10% DMSO and 4% glucose) will be administered through intradermal injection at 5 sites (100 µL/site) in the posterior cervical region, targeting lymphatic drainage into both superficial and deep cervical lymph nodes (5-10 cm from the cervical lymph nodes). Injection sites will alternate between left and right sides of the neck for each administration timepoint.
  Interventions: Biological: Tolerogenic dendritic cells (tolDC)

INTERVENTIONS:
Biological: Tolerogenic dendritic cells (tolDC) — In brief, clinical-grade tolDC vaccines will be prepared from leukapheresis starting material of non-mobilized blood and subsequent immunomagnetic selection of CD14+ monocytes using a CliniMACS device. CD14+ monocytes will then be cultured in GMP-grade cell culture medium supplemented with 2% human AB serum, GM-CSF, IL-4 and 1 alpha,25 dihydroxyvitamin D3. At day 4, tolDC will be stimulated using a cytokine cocktail to induce a migratory phenotype. At day 6, tolDC will be harvested, loaded with antigen, resuspended, and cryopreserved. Separate aliquots of the cell product are prepared for final quality control and quality assurance (QC/QA) assessment. This includes cell count, viability, phenotypic analysis using flow cytometry, and induction of T cell hyporesponsiveness in allogeneic mixed leukocyte reaction (allo-MLR).

SUMMARY:
The investigators propose to design and conduct a phase IIa clinical trial to treat patients with progressive forms of multiple sclerosis (MS) by vaccination with tolerogenic dendritic cells (tolDC), generated using Good Manufacturing Practices (GMP). Hereby, the investigators want to demonstrate the efficacy and safety of administrating clinical-grade vitamin D3-treated tolDC loaded with myelin-derived peptides to patients with progressive forms of MS. In vitro generation of dedicated and stable immunomodulatory DC followed by in vitro loading of antigens to ensure tolerance and safety of DC-directed therapy is a promising strategy with the potential to induce long term tolerance.

DETAILED DESCRIPTION:
This is an open-label, self-controlled, multi-center phase IIa clinical trial designed to evaluate the proof-of-concept for both efficacy and safety of tolDC-based therapy. The primary objective is to determine whether treatment with tolDC is effective (using a surrogate primary outcome-change in EDSS score) and safe (the occurrence and severity of adverse events). Secondary evaluations will include the clinical outcomes (assessed using 9HPT, SDMT and number and severity of relapses) and MRI-based markers. Participants will serve as their own controls, with data from 24 weeks pre-treatment period (documented by their neurologist). Following six tolDC administrations, a 24-weeks follow-period will take place. Furthermore, participants can enroll voluntarily into an optional additional follow-up phase of 52 weeks. Completion of screening assessments and confirmation of eligibility criteria should take no longer than 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years old, and ≤65 years of age, at time of screening visit
* Diagnosis of MS according to the 2017 McDonald Criteria or more recent criteria
* Progressive MS by 2014 Lublin MS phenotypic criteria
* EDSS 2,0 - ≤7,5
* No clinical evidence of relapses in the past 2 years
* Ability to understand and the willingness to sign a written informed consent document. Patients must have signed informed consent to participate in the trial.
* Appropriate venous access
* Use of adequate contraceptive measures or not of childbearing potential

Exclusion Criteria:

* Previous treatment with alemtuzumab, autologous hematopoietic stem cell transplantation or cladribine in the past 3 years.
* Prior treatment with any investigational agent within 3 months, or 5 half-lives, whichever is longer.
* Current and ongoing treatment with an approved DMT for MS
* Treatment with S1P receptor modulators, natalizumab, dimethylfumarate, teriflunomide within the last 3 months prior to study enrolment; last treatment with B cell depleting monoclonal antibodies at least 6 months prior to enrollment and normal CD19 B cell counts at time of enrollment
* Pregnancy or planning pregnancy in the next 12 months and breast feeding
* Drug or alcohol abuse
* Inability to undergo MRI assessments
* History of or actual signs of immunodeficiency or malignancies (with the exception of treated basal cell carcinoma)
* Concurrent clinically relevant cardiac, immunological, pulmonary, neurological, renal or other major disease that could impact safety or outcome measures.
* Active or chronic infection with hepatitis B, C, HIV, syphilis or tuberculosis
* Splenectomy
* Dementia or severe psychiatric, cognitive or behavioral problems or other comorbidity that could interfere with the compliance to the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy (Change in EDSS score) | 62 weeks
  To evaluate the efficacy of tolDC administration, the change in Expanded Disability Severity Scale (EDSS) will be employed. The participants' disability level well be checked during every visit. The EDSS consists of a 10-point scale of disease severity ranging from 0, i.e. no disability, to 10, i.e. death from MS.
  The impact on disability progression will be analyzed by the proportion of participants free from confirmed disability progression, defined by sustained changes in the EDSS score.
  Disease progression criteria:
  * 1.0 point in participants with a screening EDSS of 0-5.0
  * 0.5 point in those with a screening EDSS of 5.5-6.0
Incidence of treatment-emergent adverse events (safety and tolerability) | 62 weeks
  Tolerability and safety of tolDC administration will be assessed by recording the incidence, severity, and relationship to study treatment of adverse events throughout the trial.
  Participants will be monitored by the treating neurologist for the occurrence and outcomes of AEs, SAEs, relapses and study discontinuations. Full physical examinations, vital signs, and blood and urine samples (only in case of women of childbearing age for pregnancy test) will be recorded at screening, during tolDC administration and during follow-up. An assessment of severity grading of AEs will follow the WHO toxicity grading scale (1= mild, 2= moderate, 3= severe, 4= potentially life threatening).

SECONDARY OUTCOMES:
9 Hole Peg Test (9HPT) | 62 weeks
  The 9-HPT is a quantitative assessment of upper limb (arm and hand) function. The test device consists of a container containing nine pegs and a wooden or plastic board with nine empty holes. The participant is required to pick up each peg individually and place them as quickly as possible in the nine holes. Once all the pegs are placed in the holes, the participant must remove them one by one, again as quickly as possible and return them to the container. The total time to complete the task is recorded.
Symbol Digit Modalities test (SDMT) | 62 weeks
  The SDMT is a useful tool for identifying cognitive impairment as well as monitoring changes in cognitive functioning over time or in response to treatment. The SDMT is quick and easy to administer, typically taking about five minutes. The test involves a basic substitution exercise that is easily manageable for adults. Using a reference key, participants are given 90 seconds to match specific numbers with corresponding geometric figures and verbally provide their answers. A study nurse or another appropriately trained individual records the responses in writing. The final outcome is calculated by the total number of answers given minus the incorrect answers (N numbers in 90 seconds).
T2 lesion volume on MRI | 62 weeks
  T2 lesion volume on MRI scans will be evaluated to determine if administration of tolDC influences clinical and subclinical disease evolution.
Total Brain Volume on MRI | 62 weeks
  Total brain volume on MRI scans will be evaluated to determine if administration of tolDC influences clinical and subclinical disease evolution
Brain Atrophy on MRI | 62 weeks
  Atrophy rate on MRI scans will be evaluated to determine if administration of tolDC influences clinical and subclinical disease evolution
Biomarkers | 62 weeks
  Change in Neurofilament Light Chain (NfL) serum and Glial Fibirallary Acidic Protein (GFAP) serum will be assessed as biomarkers. NfL is a sensitive marker of neuroaxonal damage and has been associated with disease activity and treatment response in MS. GFAP reflects astrocytic activation and may provide insights into neuroinflammation and glial responses, particularly relevant in progressive MS. These biomarkers will be measured using ultrasensitive immunoassays, allowing for high-resolution monitoring of subclinical disease progression and treatment-related effects.
  These will be measured in serum samples and biobanked for later analysis.

OTHER OUTCOMES:
Immunological response | 62 weeks
  To comprehensively assess therapy-related immunological changes and the induction of antigen-specific tolerance, we will perform high-dimensional immune profiling using cryopreserved peripheral blood mononuclear cells (PBMCs) and matched serum/plasma samples collected at predefined time points throughout the trial. In brief, we will store samples of PBMC in biobank facilities in Antwerp and Spain prior to vaccination and during and after the IMP administrations for future centralized high-dimensional functional immune-profiling.
Patient Reported Outcomes - Visual Analog Scale (VAS) | 62 weeks
  Measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')
Patient Reported Outcomes - EuroQol 5-Dimension, 5-Level Questionnaire (EQ-5D-5L) | 62 weeks
  The EQ-5D-5L is a self-reported questionnaire designed to assess health-related quality of life. It evaluates five key dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on a five-point scale, ranging from no problems to extreme problems (e.g., I have no problems walking about, slight problems, moderate problems, severe problems or I am unable to walk). In addition to these dimensions, the questionnaire includes a VAS, where respondents rate their overall health on a scale from 0 to 100 - 0 representing the worst imaginable health and 100 the best.

CONTACTS AND LOCATIONS:
Locations (2):
- Universitair Ziekenhuis Antwerpen (UZA), Edegem, Belgium
- Germans Trias i Pujol Hospital (HUGTiP), Badalona, Spain